CLINICAL TRIAL: NCT02934087
Title: Evaluation of a Randomized Comparison of Direct Versus Snare Techniques for Cannulation of Contralateral Gate During an Endovascular Aneurysm Repair (EVAR) Procedure
Brief Title: Endovascular Aneurysm Repair (EVAR) Gate Study
Acronym: EVAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minneapolis Heart Institute Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: EV001
Record Dates: First submitted 2011-08-05; First posted 2016-10-14 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Abdominal Aortic Aneurysm (AAA)
Keywords: snare technique; cannulation of contralateral gate; endovascular; aneurysm; AAA; Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Aneurysm | interventions — Endovascular Aneurysm Repair

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Retrograde Gate Cannulation (Active Comparator): All patients undergoing elective EVAR with a standard commercially available stent graft will be randomized after informed consent obtained; gate cannulation method will be attempted for a period of 15 minutes. If unsuccessful during this time a crossover to the alternative method (snare) will be attempted. The study will be terminated at 15 minutes in the crossover arm if still unsuccessful.
  Interventions: Procedure: Endovascular Aneurysm Repair
- Snare Technique (Active Comparator): All patients undergoing elective EVAR with a standard commercially available stent graft were randomized after informed consent obtained; gate cannulation method was attempted for a period of 15 minutes. If unsuccessful during this time a crossover to the alternative method (retrograde gate cannulation) was attempted. The study will be terminated at 15 minutes in the crossover arm if still unsuccessful.
  Antegrade or crossover cannulation involves passing a guidewire from the ipsilateral limb to the contralateral limb gate of the endograft, which can be accomplished with a curved catheter. The wire may be retrieved on the contralateral limb using a snare device.
  Interventions: Procedure: Endovascular Aneurysm Repair

INTERVENTIONS:
Procedure: Endovascular Aneurysm Repair — Endovascular aneurysm repair (or endovascular aortic repair) (EVAR) is a type of endovascular surgery used to treat pathology of the aorta, most commonly an abdominal aortic aneurysm (AAA)
  Other Names: EVAR

SUMMARY:
This study will evaluate a randomized comparison of direct versus snare techniques for cannulation of contralateral gate during an endovascular aneurysm repair (EVAR) procedure.

This information will be used to determine if primary snaring is superior to retrograde cannulation in decreasing procedural time and radiation exposure.

DETAILED DESCRIPTION:
Endografts currently FDA-approved for abdominal aortic aneurysm (AAA) repair are modular systems,comprised of a main body (Aortic Trunk) and two legs (Ipsilateral Leg Endoprosthesis and a contralateral leg endoprosthesis). In placement of the endograft the main body and ipsilateral limb are deployed from a retrograde common femoral artery approach. From the contralateral femoral artery, cannulation of the contralateral gate is required to deploy the contralateral iliac limb.Cannulation of the contralateral limb gate is the portion of the operation that requires the most "wire skills." Depending on the patients' body type, angulations of the aorta and the size and volume of the AAA, this portion of the procedure can be technically difficult. This portion may become lengthy and discouraging if the surgeon fails to cannulate the gate using a particular approach. Cannulation of the contralateral limb gate from a retrograde femoral artery approach is commonly achieved by first using a maneuverable guidewire and steerable catheter. Antegrade or crossover cannulation involves passing a guidewire from the ipsilateral limb to the contralateral limb gate of the endograft, which can be accomplished with a curved catheter. The wire may be retrieved on the contralateral limb using a snare device. The problem and why it is important -- difficulty in accessing the contralateral gate leads to increase procedural time and excess exposure to radiation. The standard of care is retrograde cannulation with the use of crossover snare techniques as a secondary adjunct if retrograde cannulation fails. In this study we will compare retrograde cannulation to primary snaring.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Patient is undergoing EVAR repair with a commercially available endograft
* Willing to give consent
* Procedure is Elective

Exclusion Criteria:

* Declines to participate
* Unable to provide consent
* Urgent AAA repair
* Participating in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2011-08; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Primary Endpoint: Time to contralateral gate cannulation | Intra-operatively comparing the time to contralateral gate cannulation (snare or retrograde techniques) .
  The patient will be randomized to either a snare or retrograde technique in a 1:1 ratio intraoperatively at the time of deployment of the main body of the graft. The timer will be started at 0 when positioning catheter is withdrawn from para-renal position into sac. The timer will be stopped after successful gate cannulation or after 30 minutes of fluoroscopy time.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Titus, MD, Principal Investigator — Minneapolis Heart Institute Foundation
Locations (1):
- Minneapolis Heart Institute, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided